CLINICAL TRIAL: NCT03292445
Title: Induction of Immune Tolerance by Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T Cell Transfusion in HLA Haplotype Matched Related and 3 Antigen HLA Matched Unrelated Living Donor Kidney Transplantation
Brief Title: Inducing Graft Tolerance in HLA Haplotype Matched Related and 3 Ag Matched Unrelated Living Donor Kidney Transplantation
Acronym: CIRM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samuel Strober (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Samuel Strober, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40442
Record Dates: First submitted 2017-09-05; First posted 2017-09-25 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Immune Tolerance

STUDY DESIGN:
Intervention Model Description: Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T Cell Transfusion in HLA Haplotype Matched Related and 3 Ag HLA Matched Unrelated Living Donor Kidney Transplantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune tolerance after kidney transplant (Experimental): Immune tolerance after kidney transplant will be induced by transfusion of enriched donor blood stem cells and T cells to initiate blood cell mixed chimerism in patients conditioned with total lymphoid irradiation and rabbit anti-thymocyte globulin after kidney transplant. Patients will receive corticosteroids for 14 weeks with gradual dose reduction. They will also receive 12 months of mycophenolate mofetil and 18 months of tacrolimus with dose tapering beginning 9 months post-transplant and continuing as long as mixed chimerism is maintained and there is no evidence of graft versus host disease and no kidney rejection evident. Patients losing chimerism will continue on low dose immunosuppressive drug doses unless additional kidney rejection therapy is needed.
  Interventions: Procedure: Immune tolerance after kidney transplant; Drug: Donor blood stem cells and T cells

INTERVENTIONS:
Procedure: Immune tolerance after kidney transplant — Induction of immune tolerance after kidney and hematopoietic cell transplantation with a conditioning regimen of total lymphoid irradiation and anti-thymocyte globulin followed by immunosuppressive drugs for 18 months. Immunosuppressive drugs are stopped if stable chimerism is achieved and there is no kidney rejection.
Drug: Donor blood stem cells and T cells — Immune tolerance after kidney transplantation resulting from mixed blood cells chimerism will be induced by donor blood stem cells and T cells given to the kidney recipient. Donor cells will be collected by apheresis after "mobilization" of blood stem cells from bone marrow 6-8 weeks before kidney transplant. Collected cells will undergo CD34 selection to recover >10 million donor blood stem cells/kg of patient weight to be combined with up to 150 million donor T cells/kg for transfusion soon after kidney transplant. The IND for this study covers the infusion of donor blood stem cells.
  Other Names: Immune tolerance after kidney transplant

SUMMARY:
This research study is to determine if donor blood stem cells given after living, related, HLA antigen (Ag) haplotype match or living, unrelated donor kidney transplantation. Minimal HLA antigen matching will include matching of 2 HLA antigens that can be either HLA A, B, and /or DR. This research will change the immune system such that immunosuppressive drugs can be completely withdrawn or reduced to minimal dose without kidney rejection.

DETAILED DESCRIPTION:
The objectives of this study are to determine whether patients undergoing kidney transplants for end stage renal disease (ESRD) can be taken off immune suppression drugs given to prevent kidney rejection or can be maintained on low dose immune suppression while maintaining normal kidney function. Patients will receive blood stem cell transfusions from their donors 11 days after transplant to reduce the risk of graft rejection while tapering the post-transplant immune suppression drug regimen. Patients will be treated with total lymphoid irradiation (TLI) and rabbit anti-thymocyte globulin (rATG) followed by transfusion of enriched CD34+ hematopoietic cells containing blood stem cells and CD3+ T cells from their donors in order to induce blood cell mixed chimerism. These chimeric patients produce blood cells from both their own and their donors' blood stem cells. Donors will have blood collected by apheresis after treatment with drugs to "mobilize" blood stem cells from their bone marrow. Collection of the donor's cells will occur 6-8 weeks before kidney donation surgery. After transplant, patients will receive a 14 week course of corticosteroid therapy (e.g., Prednisolone) with gradual dose reduction. They will also receive a 12 month course of mycophenolate mofetil (MMF) with dose tapering beginning 9 months post-transplant and an 18 month course of Tacrolimus with tapering also beginning at 9 months post-transplant. Patients will be monitored for renal function, mixed blood cell chimerism, the appearance of donor specific antibodies (DSA) from their own immune cells reacting to the transplanted kidney, and evidence of rejection in any biopsies of the donor kidney after transplant. Immune suppression drug withdrawal will begin and continue as long as mixed chimerism is maintained, the patient shows no evidence of graft versus host disease (GVHD), the transplanted kidney functions well, and there is no indication of kidney rejection in biopsies. Patients not meeting these criteria will be maintained on low dose immunosuppressive drug therapy unless more extensive treatments are needed to prevent rejection. Potential candidates need to be approved for kidney transplant under this protocol and available for close follow-up post-transplant. This study, sponsored by the California Institute for Regenerative Medicine (CIRM), is being conducted in parallel with NCT01165762 sponsored by the National Institutes of Health with distinct reporting and separation of funding support for the patients enrolled under each sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adults (18 years of age) living donor renal transplant recipients at Stanford University Medical Center who have a one haplotype match donor.
2. Patients who agree to participate in the study and sign an Informed Consent.
3. Patients who have no known contraindication to administration of rabbit ATG or radiation.
4. Males and females of reproductive potential who agree to practice a reliable form of contraception for at least 24 months posttranplant.

Exclusion Criteria:

1. Previous treatment with rabbit ATG or known allergy to rabbit proteins.
2. History of malignancy with the exception of non-melanoma skin malignancies.
3. Pregnant women or nursing mothers.
4. Serological evidence of HIV, Hepatitis B or Hepatitis C infection.
5. Seronegative for Epstein-Barr virus , if donor is seropositive.
6. Leukopenia (with a white blood cell count < 3000/mm3) or thrombocytopenia (with a platelet count < 100,000/mm3)
7. Panel Reactive antibody greater then 20% or demonstration of donor specific antibody (DSA).
8. Prior organ transplantation.
9. High risk of primary kidney disease recurrence (i.e. primary FSGS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-02-14 (Actual); Primary Completion 2022-02-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Reduction of dependence on immunosuppressive drugs to prevent graft rejection. | 24 months post-transplant
  Percentage of patients able to maintain normal renal function after coming off all immunosuppressive drug therapy and percentage of patients maintaining normal renal function with only minimum effective dose immunosuppressive drug monotherapy.

SECONDARY OUTCOMES:
Incidence of rejection episodes requiring corticosteroid therapy | 24 months post-transplant
  Percentage of patients experiencing biopsy proven rejection episodes requiring corticosteroid therapy.
Incidence of graft loss. | 24 months post-transplant
  Percentage of patients experiencing loss of transplanted kidneys.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Md Strober, MD, Study Chair — Stanford University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976
- [Background] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Sarwal M, Millan MT, Shizuru JA, Lowsky R, Engleman EG, Strober S. Tolerance and withdrawal of immunosuppressive drugs in patients given kidney and hematopoietic cell transplants. Am J Transplant. 2012 May;12(5):1133-45. doi: 10.1111/j.1600-6143.2012.03992.x. Epub 2012 Mar 8. PMID 22405058
- [Background] Scandling JD, Busque S, Shizuru JA, Lowsky R, Hoppe R, Dejbakhsh-Jones S, Jensen K, Shori A, Strober JA, Lavori P, Turnbull BB, Engleman EG, Strober S. Chimerism, graft survival, and withdrawal of immunosuppressive drugs in HLA matched and mismatched patients after living donor kidney and hematopoietic cell transplantation. Am J Transplant. 2015 Mar;15(3):695-704. doi: 10.1111/ajt.13091. PMID 25693475
- [Result] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Millan MT, Shizuru JA, Hoppe RT, Lowsky R, Engleman EG, Strober S. Tolerance and chimerism after renal and hematopoietic-cell transplantation. N Engl J Med. 2008 Jan 24;358(4):362-8. doi: 10.1056/NEJMoa074191. PMID 18216356